CLINICAL TRIAL: NCT04106219
Title: A Phase 1 Study of Aurora Kinase A Inhibitor LY3295668 Erbumine as a Single Agent and in Combination in Patients With Relapsed/Refractory Neuroblastoma
Brief Title: A Study of LY3295668 Erbumine in Participants With Relapsed/Refractory Neuroblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: New Approaches to Neuroblastoma Therapy Consortium (NANT) (Unknown); Innovative Therapies for Children with Cancer in Europe (ITCC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17295; J1O-MC-JZHD (Other: Eli Lilly and Company); 2019-001042-18 (EudraCT Number); 2019-01 (Other: NANT); ITCC-085 (Other: ITCC)
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: aurora kinase A; kinase; aurora A; aurora kinase inhibitor; aurora kinase A inhibitor; kinase inhibitor; AURKA; AurA; pediatric neuroblastoma; children
MeSH Terms: conditions — Neuroblastoma; Epilepsy | interventions — LY3295668 erbumine; Topotecan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3295668 Erbumine Escalation (Experimental): LY3295668 Erbumine given orally.
  Interventions: Drug: LY3295668 Erbumine
- LY3295668 Erbumine + Topotecan + Cyclophosphamide Escalation (Experimental): LY3295668 Erbumine given orally and topotecan and cyclophosphamide given intravenously (IV).
  Interventions: Drug: LY3295668 Erbumine; Drug: Topotecan; Drug: Cyclophosphamide
- LY3295668 Erbumine Expansion (Experimental): LY3295668 Erbumine given orally.
  Interventions: Drug: LY3295668 Erbumine
- LY3295668 Erbumine + Topotecan + Cyclophosphamide Expansion (Experimental): LY3295668 Erbumine given orally and topotecan and cyclophosphamide given IV.
  Interventions: Drug: LY3295668 Erbumine; Drug: Topotecan; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: LY3295668 Erbumine — Administered orally.
Drug: Topotecan — Administered IV.
  Arms: LY3295668 Erbumine + Topotecan + Cyclophosphamide Escalation; LY3295668 Erbumine + Topotecan + Cyclophosphamide Expansion
Drug: Cyclophosphamide — Administered IV.
  Arms: LY3295668 Erbumine + Topotecan + Cyclophosphamide Escalation; LY3295668 Erbumine + Topotecan + Cyclophosphamide Expansion

SUMMARY:
The reason for this study is to see if the study drug LY3295668 erbumine is safe in participants with relapsed/refractory neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have relapsed/refractory neuroblastoma and have active disease in at least one site: bone, bone marrow or soft tissue. Participants must be able to submit an archival sample of tissue.
* Participants must be able to swallow capsules.

Exclusion Criteria:

* Participants must not have had an allogeneic hematopoietic stem cell, bone marrow, or solid organ transplant.
* Participants must not have untreated tumor that has spread to the brain or spinal cord.
* Participants must not have a serious active disease other than neuroblastoma.
* Participants must not have a condition affecting absorption.
* Participants must not have had prior aurora kinase inhibitor exposure.
* Participants must not have a known allergy to the study treatment.
* Participants must not have symptomatic human immunodeficiency virus (HIV) infection or symptomatic activated/reactivated hepatitis A, B, or C.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Baseline through Cycle 2 (28 Day Cycle)
  Number of Participants with DLTs
Overall Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR) | Baseline through Measured Progressive Disease (Estimated up to 5 Years)
  ORR
Duration of Response (DoR) | Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Estimated up to 5 Years)
  DoR

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3295668 | Cycle 1 Day 1 through Cycle 1 Day 15 (28 Day Cycles)
  PK: AUC of LY3295668
PK: AUC of LY3295668 in Combination with Topotecan and Cyclophosphamide | Cycle 1 Day 1 through Cycle 1 Day 15 (28 Day Cycles)
  PK: AUC of LY3295668 in Combination with topotecan and cyclophosphamide
Best Overall Response (BOR): Percentage of Participants with CR, PR, Stable Disease (SD), or Progressive Disease (PD) | Baseline to Date of Objective Disease Progression (Estimated up to 5 Years)
  BOR
Progression-Free Survival (PFS) | Baseline to Objective Progression or Death Due to Any Cause (Estimated up to 5 Years)
  PFS
Overall Survival (OS) | Baseline to Date of Death from Any Cause (Estimated up to 6 Years)
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (7):
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Chicago - Comer Children's Hospital, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Childrens Hospital, Houston, Texas
- Perth Children's Hospital, Perth, Western Australia, Australia
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium
- France (2):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Institut Curie, Paris
- Universitätsklinikum Köln, Cologne, Germany
- Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Infantil Universitario Niño Jesús, Madrid
- Alder Hey Children's Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3295668 Erbumine in Participants With Relapsed/Refractory Neuroblastoma — https://trials.lillytrialguide.com/en-US/trial/50gRHl2d9N02mw6yfhdI4Z